CLINICAL TRIAL: NCT04550013
Title: The Effect of Low-Load Resistance Training With Blood Flow Restriction for Treatment of Chronic Patellar Tendinopathy - A Randomized Clinical Trial
Brief Title: Blood Flow Restriction Training for Treatment of Chronic Patellar Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University College Absalon (Other); Danske Fysioterapeuter (Other)
Responsible Party: Principal Investigator, Mikkel Holm Hjortshøj Jensen, Principal Investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A2359
Record Dates: First submitted 2020-08-20; First posted 2020-09-16 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Patellar Tendinopathy; Jumper's Knee
Keywords: Patellar tendinopathy; Overuse Injury; Rehabilitation
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to intervention allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy-Slow Resistance training (Active Comparator): Heavy-Slow Resistance training. Three times weekly for 12 weeks.
  Interventions: Other: Heavy-Slow Resistance training
- Low-Load Blood Flow Restriction training (Experimental): Low-Load Blood Flow Restriction training. Three times weekly for 12 weeks
  Interventions: Other: Low-Load Blood Flow Restriction training

INTERVENTIONS:
Other: Heavy-Slow Resistance training — Resistance training for knee extensors. The exercise will be performed at 80% of 1 RM and slowly (6 s/repetition).
  Arms: Heavy-Slow Resistance training
Other: Low-Load Blood Flow Restriction training — Resistance training for knee extensors. The exercise will be performed at 30% of 1 RM and with a relative Artery Occlusion Pressure of 80%
  Arms: Low-Load Blood Flow Restriction training

SUMMARY:
The purpose of this study is to investigate the clinical and functional outcome of a 12-week rehabilitation regime consisting of Low-Load Blood Flow Restriction compared to Heavy-Slow Resistance training in male patients with chronic unilateral patellar tendinopathy.

DETAILED DESCRIPTION:
Chronic tendinopathy represents a considerable problem in both elite and recreational athletes, and symptoms may affect athletic performance and reduce or even result in retirement from sports participation. The current best treatment is considered to be heavy-slow resistance training (HSRT); however, not all patients are able to cope with heavy exercise loads. Therefore, low-load strength training performed under partial blood flow restriction may be a clinically relevant rehabilitation tool.

This project aims to investigate a new innovative intervention to treat chronic unilateral patellar tendinopathy in male individuals using strength training with low-load muscle contractions performed under partial blood flow restriction (LL-BFR), and to compare the resulting treatment outcome to that of the current best practice (HSRT). Specifically, the effect of LL-BFR will be investigated using a randomized controlled trial design with two groups; 1) a low-load blood flow restriction training program, and 2) a heavy-load slow strength training program. A total sample size of 36 participants are needed when assuming a 10 % dropout.

The training protocol consist of three weekly training sessions during a 12-week rehabilitation period. The primary outcome is measured using the Single-Leg Decline Squat at 12-week.

If LL-BFR proves to be an effective treatment strategy for tendinopathy, it can easily be implemented in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral patellar tendinopathy
* Chronic (symptoms >3 months)
* Pain of ≥ 4 during preferred sporting activity on the numerical pain rating scale (NRS; with 0 being no pain and 10 being the worst imaginable pain)
* Ultrasonographical tendon swelling
* Ultrasonographical hypo-echoic area with doppler

Exclusion Criteria:

* Bilateral tendinopathy
* Cardiovascular diseases
* Diabetes
* Smoking
* Previous surgery or trauma to the knee joint with an effect on the presenting clinical condition
* Participants must not have been enrolled in a resistance based-rehabilitation program for the affected patellar tendon within the previous three months
* Previous corticosteroid injection for patellar tendinopathy

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-09-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline - 12 weeks using the clinical functional test Single-Leg Decline Squat measured on the Numerical Rating Scale (NRS; 0= no pain, 10 = worst imaginable pain) | Baseline-12 weeks.
  Single-Leg Decline Squat is a reliable patellar tendon pain provocation test used to assess pain during function.

SECONDARY OUTCOMES:
Single-Leg Decline Squat test | Baseline, 3, 6 weeks + 1 year follow-up
  A reliable patellar tendon pain provocation test, will be used to assess pain during function using the Numerical Rating Scale (NRS; 0= no pain, 10 = worst imaginable pain)
Pain rating on Numeric Rating Scale (NRS; 0 = no pain; 10 = worst imaginable pain) during training. | Baseline, 3, 6 and 12 weeks + 1 year follow-up
Self-reported activity level of sporting activities (hours/week) | Baseline, 3, 6 and 12 weeks + 1 year follow-up
  Participants will self-report how many hours a week they are performing sporting activities: We will monitor to see if they decrease, maintain or increase hours per week of sporting activity
Doppler activity using Ultrasonography power Doppler | Baseline, 3, 6 and 12 weeks + 1 year follow-up
  Using Ultrasonography, we will measure Doppler activity within the affected tendon and use ImageJ for the analysis
Tendon thickness measured using Ultrasonography | Baseline, 3, 6 and 12 weeks + 1 year follow-up
Muscle cross-sectional area measured using Ultrasonography | Baseline, 3, 6 and 12 weeks + 1 year follow-up
  We will measure the muscle thickness of vastus lateralis using ultrasonography
Muscle structure measured by MRI | Baseline and 12 weeks
Tendon dimensions measured by MRI | Baseline and 12 weeks
Isometric Muscle Strength | Baseline, 3, 6 and 12 weeks + 1 year follow-up
  Maximal muscle strength of the knee extensors is obtained during a maximal isometric voluntary contractions
Pain Pressure Threshold | Baseline, 3, 6 and 12 weeks + 1 year follow-up
  Measured by a handheld pressure algometry at most painful site, Apex Patellar, Tibialis Anterior and Extensor Carpi Radialis.
Adverse events | Baseline-12 weeks + 1 year follow-up
  Participants will self-report adverse events during intervention period and at 1 year follow-up
Victorian Institute of Sports Assessment - Patellar Tendinopathy | Baseline, 3, 6 and 12 weeks + 1 year follow-up
  The VISA-P is a questionnaire that assesses symptoms, simple test of function, and the ability to play sports. Max score for asymptomatic is 100 and worst score is 0

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Holm Hjortshøj Jensen, MSc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Physical and Occupational Therapy / Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hjortshoej MH, Juneja H, Svensson RB, Herzog RB, Lundgaard-Nielsen M, Nielsen FK, Wulff MW, Olsen AE, Nybing JD, Hansen P, Petersen J, Kjaer M, Aagaard P, Magnusson SP, Couppe C. Effect of Low-Load Blood-Flow Restricted Training Versus Heavy Slow Resistance Training in Unilateral Patellar Tendinopathy: A Randomized Clinical Trial. Scand J Med Sci Sports. 2025 Dec;35(12):e70186. doi: 10.1111/sms.70186. PMID 41452311